CLINICAL TRIAL: NCT00687999
Title: Non-insulin-dependent Diabetes Mellitus and Insulin Resistance in Chronic Hepatitis C Patients Treated With Combination Therapy With Pegylated Interferon and Ribavirin in Taiwan
Brief Title: NIDDM and IR in Combination Therapy for CHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Wan-Long Chuang, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-940055
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Hepatitis C; Insulin Resistance
Keywords: Chronic hepatitis C; diabetes; Insulin resistance; combination therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance; Diabetes Mellitus | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: pegylated interferon alpha and ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha and ribavirin — standard pegylated interferon alpha and ribavirin
  Other Names: PEG-IFN-alpha

SUMMARY:
The influence of insulin sensitivity and glucose tolerance on the effects of antiviral therapy for HCV remains unclear. The aim of the present study was (1) To elucidate the clinical and virological factors associated with sustained viral response in patients with combination therapy with PEG-IFN and ribavirin. (2) To clarify the influence of diabetes mellitus (DM), impaired glucose tolerance test (IGT) and insulin resistance (IR) on the HCV response to combination therapy with PEG-IFN and ribavirin. (3) To test the influence of combination therapy on HOMA IR

DETAILED DESCRIPTION:
Total 300 treatment-naïve chronic hepatitis C patients will be enrolled. The prevalence of NIDDM, IGT and IR will be explored in this hospital-based study among the clinically defined chronic hepatitis C Taiwanese. The clinical manifestations of chronic hepatitis C in the biochemical, virological and histopathological aspects will be evaluated. Liver enzymes will be measured on a multichannel autoanalyzer. Virological markers for HCV including serum HCV RNA detected using a standardized automated qualitative PCR assay, HCV RNA genotypes determined for genotypes 1a, 1b, 2a, 2b and 3a and serum HCV RNA levels measured by using the branched DNA assay. The liver histology will be assessed for scoring the disease activity grade quantitatively according to the histological activity index (HAI). Patients are assigned a diagnosis of DM if there was documented use of oral hypoglycemic medication or insulin, random glucose in excess of 200 mg/dL, or fasting glucose greater than 126 mg/dL on two occasions. A standard oral glucose tolerance test (OGTT) will be performed. In addition to an OGTT, a history of diabetes mellitus by chart review and/or questionnaire will be also obtained. Standard antiviral therapy will be carried out with PEG-IFN, given subcutaneously weekly plus 1,000-1,200 mg of oral ribavirin daily. Patients will receive another 24 week of follow-up period to determine the virological response.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis C patients with positive anti-HCV for more than 6 months and HCV RNA
2. No overt hepatic failure or decompensated liver cirrhosis (Child-Pugh class B or C) or hepatocellular carcinoma.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen (HBsAg)or with concomitant human immunodeficiency virus infection
2. With other types of hepatitis including autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, Wilson's disease, alpha 1-antitrypsin deficiency
3. Current or past history of alcohol abuse (80 mL ethanol per day)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) rate, HCV RNA seronegative by PCR throughout 24-week off-treatment period; biochemical, virological and histological characteristics of CHC patients; HOMA-IR change after combination therapy | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Long Chuang, MD, PhD., Principal Investigator — Department of Internal Medicine, Kaohsiung Medical University Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Mason AL, Lau JY, Hoang N, Qian K, Alexander GJ, Xu L, Guo L, Jacob S, Regenstein FG, Zimmerman R, Everhart JE, Wasserfall C, Maclaren NK, Perrillo RP. Association of diabetes mellitus and chronic hepatitis C virus infection. Hepatology. 1999 Feb;29(2):328-33. doi: 10.1002/hep.510290235. PMID 9918906
- [Background] Shintani Y, Fujie H, Miyoshi H, Tsutsumi T, Tsukamoto K, Kimura S, Moriya K, Koike K. Hepatitis C virus infection and diabetes: direct involvement of the virus in the development of insulin resistance. Gastroenterology. 2004 Mar;126(3):840-8. doi: 10.1053/j.gastro.2003.11.056. PMID 14988838
- [Background] Lecube A, Hernandez C, Simo R, Esteban JI, Genesca J. Glucose abnormalities are an independent risk factor for nonresponse to antiviral treatment in chronic hepatitis C. Am J Gastroenterol. 2007 Oct;102(10):2189-95. doi: 10.1111/j.1572-0241.2007.01402.x. Epub 2007 Jul 7. PMID 17617205
- [Background] Lee SD, Yu ML, Cheng PN, Lai MY, Chao YC, Hwang SJ, Chang WY, Chang TT, Hsieh TY, Liu CJ, Chen DS. Comparison of a 6-month course peginterferon alpha-2b plus ribavirin and interferon alpha-2b plus ribavirin in treating Chinese patients with chronic hepatitis C in Taiwan. J Viral Hepat. 2005 May;12(3):283-91. doi: 10.1111/j.1365-2893.2005.00590.x. PMID 15850469
- [Background] Romero-Gomez M, Del Mar Viloria M, Andrade RJ, Salmeron J, Diago M, Fernandez-Rodriguez CM, Corpas R, Cruz M, Grande L, Vazquez L, Munoz-De-Rueda P, Lopez-Serrano P, Gila A, Gutierrez ML, Perez C, Ruiz-Extremera A, Suarez E, Castillo J. Insulin resistance impairs sustained response rate to peginterferon plus ribavirin in chronic hepatitis C patients. Gastroenterology. 2005 Mar;128(3):636-41. doi: 10.1053/j.gastro.2004.12.049. PMID 15765399
- [Background] D'Souza R, Sabin CA, Foster GR. Insulin resistance plays a significant role in liver fibrosis in chronic hepatitis C and in the response to antiviral therapy. Am J Gastroenterol. 2005 Jul;100(7):1509-15. doi: 10.1111/j.1572-0241.2005.41403.x. PMID 15984973